CLINICAL TRIAL: NCT06244654
Title: Anxiolytic Effectiveness of Virtual Reality Glasses in Upper Extremity Surgery
Brief Title: Anxiolytic Effectiveness of Virtual Reality Glasses in Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Burak NALBANT, assistant professor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E2-23-4787
Record Dates: First submitted 2024-01-19; First posted 2024-02-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Anesthesia; Anxiety; Postoperative Pain; Postoperative Recovery
MeSH Terms: conditions — Anxiety Disorders; Pain, Postoperative | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standart Anesthesia management (Other): In the non-VR group, the standard anesthesia procedure will be followed. Brachial plexus nerve block will be performed with a 50mm peripheral block needle (Vygon echoplex+ 22Gx50mm) with a mixture of 2% lidocaine and 0.5% bupivacaine (10 mL each) prepared as 20ml. After waiting for a sufficient time, the nerve block effectiveness of the patients will be measured by Modified Broomage scale and pinprick. Additional sedative agents may be applied to both groups at the discretion of the anesthesiologist and will be recorded. Anesthesia management will be applied to both groups in accordance with the standard working order of the Anesthesia clinic.
  Interventions: Other: No VR
- VR group (Experimental): Oculus Quest 2 VR virtual reality glasses and wired over-ear headphones will be used for patients to hear the sounds of the immersive environment and to block the sounds coming from the operating room environment. Brachial plexus nerve block will be performed with a 50mm peripheral block needle (Vygon echoplex+ 22Gx50mm) with a mixture of 2% lidocaine and 0.5% bupivacaine (10 mL each) prepared as 20ml. After waiting for a sufficient time, the nerve block effectiveness of the patients will be measured by Modified Broomage scale and pinprick.Additional sedative agents may be applied to both groups at the discretion of the anesthesiologist and will be recorded. Anesthesia management will be applied to both groups in accordance with the standard working order of the Anesthesia clinic.
  Interventions: Device: Oculus Quest 2 VR virtual reality glasses and wired over-ear headphones

INTERVENTIONS:
Device: Oculus Quest 2 VR virtual reality glasses and wired over-ear headphones — After the VR group comes to the preoperative area and is evaluated, they will be asked to wear VR glasses and headphones. VR glasses and headphones were worn on the patient during peripheral nerve block applications and the operation. At the end of the operation, the VR glasses and headphones were removed and they were taken to the postoperative recovery room.
  Arms: VR group
Other: No VR — After evaluation of the patients taken to the preoperative area, routine peripheral nerve block application was performed without the use of VR glasses. VR glasses were not worn during the operation, as is the routine protocol. At the end of the surgery, they were taken to the postoperative recovery room.
  Other Names: Control group
  Arms: Standart Anesthesia management

SUMMARY:
Regional anesthesia allows surgery without affecting the patient's level of consciousness.However, this may cause anxiety in some patients.In previous research, scientists have tried to prevent anxiety with non-pharmacological interventions such as music and cognitive therapies.Virtual reality is thought to offer an immersive experience that can alter the mind's perception of pain. Scientists have found in previous preliminary studies that virtual reality is safe and effective as an adjunct to standard sedative/analgesic protocols for reducing patients' pain and anxiety during endoscopy, colonoscopy, dental treatments, burn dressings, and labor. In this study, it is expected that anxiety scores, postoperative analgesic need and intraoperative sedation need will decrease, recovery quality will improve and patient satisfaction will increase in patients who will undergo upper extremity surgery under regional anesthesia and watch videos through VR glasses.

ELIGIBILITY:
Inclusion Criteria:

* who will undergo upper extremity surgery under regional anesthesia

Exclusion Criteria:

* being under 18 years old
* Those who do not have the ability to read, understand and sign the consent form
* An active infection or open wound in the face or eye area
* History of seizures due to an epileptic condition or any other reason
* Planning to wear a hearing aid during the surgical procedure
* Having a pacemaker or other implanted medical device
* Migraine
* Having an infectious condition that is transmitted through droplets or airborne
* not knowing Turkish
* Not deemed suitable for the approach by the surgeon
* History of psychosis or claustrophobia
* Being visually and/or hearing impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2024-01-25 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Scale | Preoperative, Postoperative 4.hour
  preoperative and postoperative STAI I and II score questions will be asked.

SECONDARY OUTCOMES:
systolic blood pressure | Preoperative, İntraoperative 0 min, İntraoperative 60min, End of Operation, Postoperative 4.hour
  non invasive systolic blood pressure measurement
diastolic blood pressure | Preoperative, İntraoperative 0 min, İntraoperative 60min, End of Operation, Postoperative 4.hour
  non invasive diastolic blood pressure measurement
mean arterial pressure | Preoperative, İntraoperative 0 min, İntraoperative 60min, End of Operation, Postoperative 4.hour
  mean blood pressure measurement
heart rate | Preoperative, İntraoperative 0 min, İntraoperative 60min, End of Operation, Postoperative 4.hour
  intraoperatif and perioperatif ecg monitarization
oxygen saturation | Preoperative, İntraoperative 0 min, İntraoperative 60min, End of Operation, Postoperative 4.hour
  intraoperatif and perioperative pulse oxymeter measurement
aditional analgesic requirement | postoperative up to 24 hour
  postoperative additional analgesic requirement
VAS score | Postoperative 1.hour, 4.hour., 12.hour., 24hour.
  A blinded evaluator will evaluate the visual analog scale score.
Patient satisfaction scale | Postoperative 4.hour
  A blinded evaluator will evaluate the Patient satisfaction scale
Surgeon satisfaction scale | Postoperativ 1.hour
  A blinded evaluator will evaluate the surgeon satisfaction scale
The quality of recovery-15 (QoR-15) | Preoperative, Postoperative 24.hour
  A blinded evaluator will evaluate the QoR-15 scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moon JY, Shin J, Chung J, Ji SH, Ro S, Kim WH. Virtual Reality Distraction during Endoscopic Urologic Surgery under Spinal Anesthesia: A Randomized Controlled Trial. J Clin Med. 2018 Dec 20;8(1):2. doi: 10.3390/jcm8010002. PMID 30577461
- [Background] Barry KS, Nimma SR, Spaulding AC, Wilke BK, Torp KD, Ledford CK. Perioperative Outcomes of Immersive Virtual Reality as Adjunct Anesthesia in Primary Total Hip and Knee Arthroplasty. Arthroplast Today. 2022 Oct 22;18:84-88. doi: 10.1016/j.artd.2022.09.015. eCollection 2022 Dec. PMID 36312886
- [Background] Alaterre C, Duceau B, Sung Tsai E, Zriouel S, Bonnet F, Lescot T, Verdonk F. Virtual Reality for PEripheral Regional Anesthesia (VR-PERLA Study). J Clin Med. 2020 Jan 13;9(1):215. doi: 10.3390/jcm9010215. PMID 31941129